Title: The Effect of Oral Guaifenesin on Pediatric Chronic Rhinitis: A Pilot Study

NCT #: NCT01364467

Document approval date: February 25, 2019

Document Type: Statistical Analysis Plan

## Statistical Analysis

Data were logged into Excel spreadsheets and analyzed by StatView 5.0 (SAS, Cary, NC). Subject demographic were compared among groups using the t test for continuous variables and the chi squared test for proportions. Significance was defined as P<0.05.